CLINICAL TRIAL: NCT00554242
Title: Chronic Study of the Effect of Grape Seed Extract Plus Ascorbic Acid on Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Effect of Grape Seed Extract Plus Ascorbic Acid on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Joseph A. Vita, MD, Boston University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-26356
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease
Keywords: endothelium; antioxidants; flavonoids
MeSH Terms: conditions — Coronary Artery Disease | interventions — Grape Seed Extract; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Grape seed extract and ascorbic acid — Grape seed extract 450 mg and ascorbic acid 1500 mg daily

SUMMARY:
A pilot study of 15 subjects will be conducted to confirm an acute effect of grape seed extract on endothelial function. We then will perform a a randomized, double blind, placebo controlled crossover study designed to investigate the benefit of grape seed extract/vitamin C treatment on endothelial function. Participants (n=40) will take a food supplement containing 450 mg of grape seed extract and 1500 mg of vitamin C or matching placebo for four weeks and then cross over to the alternative treatment (active supplement or placebo) for four weeks. We will examine endothelial function before and after each of the two treatment periods. The study will provide information about the vascular effects of these compounds.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* Pregnancy
* Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, gastrointestinal disorders that may impair absorption, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
* Treatment with an investigational new drug within the last 30 days.
* History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Vitamin E, Vitamin C, and beta carotene, lipoic acid, and other food or herbal supplements within 1 month of enrollment.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 1 month

SECONDARY OUTCOMES:
Fingertip Pulse Amplitude Tonometry | 1 month
Carotid-femoral pulse wave velocity | 1 month
Serum markers of inflammation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States